CLINICAL TRIAL: NCT03264105
Title: Retention Rate of Hydroxyapatite Nano-Fiber Reinforced Flowable Composite Versus Conventional Resin-Based Flowable Composite in Initially Demineralized Pits and Fissure: A One Year, Randomized Clinical Trial
Brief Title: Retention Rate of Hydroxyapatite Nano-Fiber Reinforced Flowable Composite Versus Conventional
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, safinaz hussien fahmy hassan, dental resident, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEBC-CU-2017-07-31
Record Dates: First submitted 2017-07-30; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Retention Rate of Flowable Composite in Demenerlized Pits and Fissure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary assessors will not be blind to intervention/control material due to different in material shade. However, the other assessors will be blind from the type of material they will evaluate the retention rate of the restoration; it will not be allowed amongst the assessor to exchange any information throughout the entire study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NovaPro™ Flow (Experimental): NovaPro™ Flow Flowable Composite, Nanova Biomaterials company, USA
  Interventions: Other: Hydroxyapatite Nanofiber reinforced flowable composite; Other: conventional resin-based flowable composite
- Conventional resin-based flowable composite (Active Comparator): Filtek™Supreme Ultra Flowable Restorative, 3M ESPE company, USA
  Interventions: Other: Hydroxyapatite Nanofiber reinforced flowable composite; Other: conventional resin-based flowable composite

INTERVENTIONS:
Other: Hydroxyapatite Nanofiber reinforced flowable composite — retention rate evaluation of Hydroxyapatite Nanofiber reinforced flowable composite
Other: conventional resin-based flowable composite — retention rate evaluation of conventional resin-based flowable composite

SUMMARY:
Pits and fissures have been considered as the single most important feature leading to the development of occlusal caries; About 90 % of carious lesions are found in the pits and fissures of permanent posterior teeth .Several materials and techniques have been developed to enhance the longevity of pit-and-fissure sealants, including the use of flowable composite resins as pit-and-fissure sealants

DETAILED DESCRIPTION:
Pits and fissures have been considered as the single most important feature leading to the development of occlusal caries; About 90 % of carious lesions are found in the pits and fissures of permanent posterior teeth . The complex morphology of occlusal pits and fissures makes them an ideal site for retention of bacteria and food remnants, rendering the performance of proper hygiene difficult or even impossible .

Several materials and techniques have been developed to enhance the longevity of pit-and-fissure sealants, including the use of flowable composite resins as pit-and-fissure sealants . However, the clinical longevity of flowable composite as fissure sealants is directly related to their retention, where the percentage of rate of retention differ on a 12-month follow-up examination were the partial loss rate of flowable composite material ranges from 15.5% to 16.5% and total loss were ranged from 12.7% to 13%, while on a 24-month follow-up examination the partial loss rate ranged from 18.1% to 20% and total loss rate ranged from 15.6% to 17%, and that depends on morphology of pits and fissures, adequate isolation, conditioning of enamel, application techniques, particular material characteristics like viscosity, surface tension, adequate adhesion and penetration of the material into the previously etched system of fissures.

In order to overcome the shortcomings of traditional dental composites, nanofibers or nanotubes fillers are broadly used in the academia and industry. The type of Nanofibers and Nanotubes used to reinforce dental resin composites include polymeric nanofibers, metallic nanofibers, and inorganic hydroxyapatide (HAP) nanofibers. The Hydroxyapatite Nanofibers are calcium phosphates fillers that allow the release of mineral from dental resin composite. Also HAP nanofibers possessing sufficiently high slenderness ratios and relatively long and thin structure, and create a lot of bonding points in the interface with polymeric matrix. When the composites suffer from huge pressure this allow tremendous stress transfer from weak polymeric matrix to tough HAP nanofibers; and consequently increase the mechanical properties of resin composite. So this study will examine the effect of adding HAP nanofibers on the clinical performances and retention rate of flowable resin composite.

ELIGIBILITY:
Inclusion Criteria:

Patients should be over 18 Years old. Patient should have good oral hygiene and general health. Patient with at least 2 non-cavitated initial occlusal carious lesion in first and/or second molar teeth in each quadrant of maxilla or mandible.

Exclusion Criteria:

Known allergy to any of the resins used. Clinically detectable cavitated carious lesion. Previously placed sealants or restorations. Bruxism or malocclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
retention rate evaluation of both restoration | 12 months
  restoration will be evaluated after 12 months by two investegators who ar blinded for the material used for the restoration.Each restoration will be independently evaluated using a mirror, blunt explorer, and air stream as the follows: Full retention (FR): the materials were fully present on the occlusal surfaces. Partially lost (PL): the materials were present, but as a result of either wear or loss of the material, part of a previously sealed pit or fissure, or both, was exposed.
  Totally lost (TL): no trace of materials was detected on the surface.

IPD SHARING:
Plan to Share IPD: Undecided